CLINICAL TRIAL: NCT01137383
Title: Safety and Efficacy of Locally Manufactured Pegylated Interferon in Hepatitis C Patients
Brief Title: Pegaferon and Ribavirin for Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Pars No Tarkib Co (Unknown)
Responsible Party: Shahin Merat, Tehran University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDRC.86.90
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: Pegaferon (pegylated interferon alpha 2a) + ribavirin

INTERVENTIONS:
Drug: Pegaferon (pegylated interferon alpha 2a) + ribavirin — pegylated interferon 180 micrograms subcutaneously weekly - ribavirin (oral, in two divided daily doses) 800 mg for genotype 2 and 3, 1000 or 1200mg (weight less than or greater than 75kg) for genotypes 1 and 4 - Duration: 24 weeks for genotype 2 and 3, 48 weeks for genotypes 1 and 4
  Other Names: Pegaferon

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a locally produced 40KD pegylated interferon alpha-2a (Pegaferon) in patients with hepatitis C. 100 patients will be treated using standard guidelines for hepatitis C. Response to treatment and side effects will be recorded.

DETAILED DESCRIPTION:
The product is locally produced and needs to be evaluated in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C
* Age between 15 and 65

Exclusion Criteria:

* previous treatment for chronic hepatitis C
* co-infection with human immunodeficiency virus or hepatitis B virus
* major thalassemia or hemophilia
* active drug user
* being treated for major depression or psychosis
* decompensated cirrhosis
* serum creatinine > 1.5 mg/dL
* solid organ transplant
* untreated thyroid disease
* uncontrolled diabetes mellitus
* uncontrolled autoimmune disease
* advanced cardiac or pulmonary disease.
* planning to become pregnant in the next 1.5 years
* patients with inadequate contraception
* not consenting to the study

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Sustained viral response | 6 months after end of treatment
  Negative hepatitis C viral RNA with a highly sensitive assay 6 months after end of treatment

SECONDARY OUTCOMES:
Adverse drug events | 18 months from start of treatment
  Any adverse event reported by patient or seen in laboratory data

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, MD, Study Chair — Tehran University of Medical Sciences
Locations (2):
- Iran (2):
  - Emam Hospital, Tehran
  - Shariati Hospital, Tehran

REFERENCES:
- [Derived] Jabbari H, Bayatian A, Sharifi AH, Zaer-Rezaee H, Fakharzadeh E, Asadi R, Zamini H, Shahzamani K, Merat S, Nassiri-Toosi M. Safety and efficacy of locally manufactured pegylated interferon in hepatitis C patients. Arch Iran Med. 2010 Jul;13(4):306-12. PMID 20597564